CLINICAL TRIAL: NCT03267381
Title: Circulating Blood Profile to Predict Recurrence and Response to Systemic Therapy
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Wren Laboratories LLC (Industry)
Responsible Party: Principal Investigator, Rondi Kauffmann, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC MEL 1783
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1a: Stage III melanoma diagnosis (biopsy-proven lymph node positive (this is either clinically palpable or enlarged nodes detected by imaging, which are then biopsied and have macroscopic disease).
  Interventions: Other: Blood draw (before surgery); Other: Blood draw (every 3 months)
- Arm 1b: Stage III after sentinel node biopsy (microscopic disease diagnosed on sentinel node biopsy).
  Interventions: Other: Blood draw (before surgery); Other: Blood draw (every 3 months)
- Arm 2: Stage IV- will need to stratify by current treatment with immunotherapy, targeted therapy, none
  Interventions: Other: Blood draw (before surgery); Other: Blood draw (at diagnosis)

INTERVENTIONS:
Other: Blood draw (before surgery) — Blood will be drawn before surgery
Other: Blood draw (every 3 months) — Blood will be drawn every 3 months
  Groups: Arm 1a; Arm 1b
Other: Blood draw (at diagnosis) — Blood will be drawn at time of diagnosis
  Groups: Arm 2

SUMMARY:
To study if a targeted gene expression profile of RNA, similar to the NETest, can be isolated from the peripheral blood of patients with melanoma, to identify active disease, provide an assessment of treatment responses, or predict risk of relapse, in conjunction with standard clinical assessment and imaging.

DETAILED DESCRIPTION:
* Evaluate the diagnostic efficacy of a circulating melanoma gene signature in pathologically verified Stage III melanoma at diagnosis (biopsy-proven lymph node positive) and compare this to LDH as a biomarker.
* Evaluate the diagnostic efficacy of a circulating melanoma gene signature in pathologically verified Stage IV melanoma (including pre-surgery patients as well as those on either targeted or immunotherapy) and compare this to LDH as a biomarker.
* Define the assay metrics for sensitivity and specificity in diagnosis in Stage III and IV tumors.
* Monitor molecular signature levels in blood to assess efficacy of this tool as compared to imaging or other biomarkers to define disease progression or treatment responses in Stage III and IV treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Primary melanoma > 1 mm in Breslow depth
3. Stage III or IV disease as determined either by sentinel node biopsy, biopsy of clinically enlarged lymph nodes, and/or imaging. If stage IV, must have tissue biopsy confirming presence of stage IV melanoma

Exclusion Criteria:

1. Pregnant patients
2. Contraindication to contrasted imaging (due to allergy or renal insufficiency)
3. Serum PCV <30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of stage III or IV melanoma.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Efficacy (stage III) | Up to 24 months
  Evaluate the diagnostic efficacy of a circulating melanoma gene signature in pathologically verified Stage III melanoma at diagnosis (biopsy-proven lymph node positive) and compare this to LDH as a biomarker.
Assay Metrics | Up to 24 months
  Define the assay metrics for sensitivity and specificity in diagnosis in Stage III and IV tumors.
Molecular signature levels | Up to 24 months
  Monitor molecular signature levels in blood to assess efficacy of this tool as compared to imaging or other biomarkers to define disease progression or treatment responses in Stage III and IV treated patients.
Efficacy (Stage IV) | Up to 24 months
  Evaluate the diagnostic efficacy of a circulating melanoma gene signature in pathologically verified Stage IV melanoma (including pre-surgery patients as well as those on either targeted or immunotherapy) and compare this to LDH as a biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Rondi Kauffmann, MD, Principal Investigator — vanderbilt Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States